CLINICAL TRIAL: NCT04790227
Title: MRI for Response Evaluation After Chemoradiation for Locally Advanced Rectal Cancer
Brief Title: MRI for Selection of Complete Responders After Chemoradiation for Locally Advanced Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Yehia Hefz Abd El.wanis, Resident, Assiut University
Other Study IDs: MRI Rectum
Record Dates: First submitted 2020-05-04; First posted 2021-03-10 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Cancer, Rectum
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — MRI

SUMMARY:
The purpose of our study is to evaluate the accuracy of MRI for selection of complete responders after chemoradiation for locally advanced rectal cancer .

DETAILED DESCRIPTION:
The current standard of care for patients with T3 or T4 and/or node-positive rectal adenocarcinoma is to offer preoperative concomitant chemoradiotherapy(CRT) followed by total mesorectal excision (TME). 1 In 10-24% of patients, no residual tumor is found at histology after surgery.2 These complete responders are known to have a very good prognosis, in terms of overall and disease-free survival.2 A complete response also raises the hotly debated question of whether surgery is still necessary for these patients, especially because total mesorectal excision (TME) may have associated morbidity and even mortality and has the potential risk of a permanent colostomy.

Recently, a more conservative treatment is advocated in patients who show a good or complete response to neoadjuvant treatment. In 2006, Habr-Gama et al. Presented the long-term results of a prospective trial that investigated a "wait-and-see" policy in a carefully selected group of patients with clinical and radiological evidence of a complete response after neoadjuvant CRT. Results at 5-year follow-up were favorable for the nonsurgical group, with an overall and disease-free survival of 93% and 85%, respectively 3.

Recently, A watch and wait policy avoids the morbidity associated with radical surgery and preserves oncologic outcomes. It could be considered a therapeutic option in patients with locally advanced rectal cancer following chemoradiotherapy with a complete clinical response.4 To safely omit surgery, it is essential to select accurately the right candidates, i.e., the true complete responders. This selection is mainly performed using digital examination, endoscopy, and biopsy, but these methods are not infallible.

High-resolution magnetic resonance imaging (MRI) has been used to assess tumor response before surgical resection. By applying the principals of histopathologic TRG and by exploiting the characteristic MRI low-signal-intensity appearances of fibrosis, it has been possible to develop a similar MRI-based TRG system. The MRI-assessed TRG (mrTRG) was found to be an independent prognostic factor for overall survival (OS) and DFS.5 Complete pathologic response (pCR) after CRT has led to the proposal of a nonoperative approach as an alternate treatment for highly selected patients with a complete clinical response (CR). Habr-Gama et al reported findings from 99 patients with a clinical CR who were treated with observation alone. The 5-year OS and DFS rates were 93% and 85%, respectively.6 In a recent study, MRI-assessed complete tumor response was strongly correlated with pathologic complete response and, therefore, can be used as a surrogate marker to predict absence of viable tumor cells.7 Recently, Diffusion-weighted MRI (DWI) could be useful for response evaluation after chemoradiation treatment (8-10) In 2009, Kim et al. showed in a study of 40 patients that DWI in addition to standard MRI significantly improved the performance of radiologists to select complete responders compared with standard MRI only

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old with locally advanced rectal adenocarcinoma (T3c-T4 N any, CRM+ M0) treated with neoadjuvant chemoradiotherapy

  * Baseline and post treatment MRI scans required for each patient;
  * Clinical assessment including digital rectal examination, and endoscopy are needed for each patient

Exclusion Criteria:

* - Patient who is not fit for preoperative CRT

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 18 years old with locally advanced rectal adenocarcinoma (T3c-T4 N any, CRM+ M0) treated with neoadjuvant chemoradiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
MRI for selection of chemoradiation response evaluation for cancer rectum | Baseline
  The purpose of our study is to evaluate the accuracy of MRI for response evaluation
  after chemoradiation for locally advanced rectal cancer . Primary outcome includes Tumor site, size, volume, extension, T2, DWI signal intensity.
  Secondary outcome after chemo-radiotherapy in T2, DWI signal intensity changes
Secondary outcome after chemo-radiotherapy | 2 months
  in T2, DWI signal intensity changes T2, DWI signal intensity changes

CONTACTS AND LOCATIONS:
Overall Officials: Shymaa Abdallah, Lecturer, Study Director — Assiut University; Hossam Eldin Galal, Proffesor, Study Chair — Assiut University
Locations (1):
- Assuit University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maas M, Nelemans PJ, Valentini V, Das P, Rodel C, Kuo LJ, Calvo FA, Garcia-Aguilar J, Glynne-Jones R, Haustermans K, Mohiuddin M, Pucciarelli S, Small W Jr, Suarez J, Theodoropoulos G, Biondo S, Beets-Tan RG, Beets GL. Long-term outcome in patients with a pathological complete response after chemoradiation for rectal cancer: a pooled analysis of individual patient data. Lancet Oncol. 2010 Sep;11(9):835-44. doi: 10.1016/S1470-2045(10)70172-8. Epub 2010 Aug 6. PMID 20692872
- [Background] Habr-Gama A, Perez RO, Proscurshim I, Campos FG, Nadalin W, Kiss D, Gama-Rodrigues J. Patterns of failure and survival for nonoperative treatment of stage c0 distal rectal cancer following neoadjuvant chemoradiation therapy. J Gastrointest Surg. 2006 Dec;10(10):1319-28; discussion 1328-9. doi: 10.1016/j.gassur.2006.09.005. PMID 17175450
- [Background] On J, Aly EH. 'Watch and wait' in rectal cancer: summary of the current evidence. Int J Colorectal Dis. 2018 Sep;33(9):1159-1168. doi: 10.1007/s00384-018-3116-5. Epub 2018 Jul 5. PMID 29978363
- [Background] Patel UB, Taylor F, Blomqvist L, George C, Evans H, Tekkis P, Quirke P, Sebag-Montefiore D, Moran B, Heald R, Guthrie A, Bees N, Swift I, Pennert K, Brown G. Magnetic resonance imaging-detected tumor response for locally advanced rectal cancer predicts survival outcomes: MERCURY experience. J Clin Oncol. 2011 Oct 1;29(28):3753-60. doi: 10.1200/JCO.2011.34.9068. Epub 2011 Aug 29. PMID 21876084
- [Background] Fayaz MS, Demian GA, Fathallah WM, Eissa HE, El-Sherify MS, Abozlouf S, George T, Samir SM. Significance of Magnetic Resonance Imaging-Assessed Tumor Response for Locally Advanced Rectal Cancer Treated With Preoperative Long-Course Chemoradiation. J Glob Oncol. 2016 Feb 10;2(4):216-221. doi: 10.1200/JGO.2015.001479. eCollection 2016 Aug. PMID 28717704
- [Background] Kim SH, Lee JM, Hong SH, Kim GH, Lee JY, Han JK, Choi BI. Locally advanced rectal cancer: added value of diffusion-weighted MR imaging in the evaluation of tumor response to neoadjuvant chemo- and radiation therapy. Radiology. 2009 Oct;253(1):116-25. doi: 10.1148/radiol.2532090027. PMID 19789256
- [Background] Sun YS, Zhang XP, Tang L, Ji JF, Gu J, Cai Y, Zhang XY. Locally advanced rectal carcinoma treated with preoperative chemotherapy and radiation therapy: preliminary analysis of diffusion-weighted MR imaging for early detection of tumor histopathologic downstaging. Radiology. 2010 Jan;254(1):170-8. doi: 10.1148/radiol.2541082230. Epub 2009 Dec 17. PMID 20019139
- [Background] Kremser C, Judmaier W, Hein P, Griebel J, Lukas P, de Vries A. Preliminary results on the influence of chemoradiation on apparent diffusion coefficients of primary rectal carcinoma measured by magnetic resonance imaging. Strahlenther Onkol. 2003 Sep;179(9):641-9. doi: 10.1007/s00066-003-1045-9. PMID 14628131